CLINICAL TRIAL: NCT03346993
Title: Can Latency of Action in Infraclavicular Brachial Plexus Block be Shortened With Warmed Bupivacaine?
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Erzurum Palandöken State Hospital (Other Government)
Responsible Party: Principal Investigator, Erkan Cem ÇELİK, Consult of Anesthesiologhy, Erzurum Palandöken State Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Palandöken State Hospital
Record Dates: First submitted 2017-11-08; First posted 2017-11-20 (Actual); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Effect Increased
Keywords: Bupivacaine; Brachial Plexus Block; Ultrasound
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 24C° 0,5% bupivacaine group (Experimental): 24C° 0,5% bupivacaine group will be performed USG guided infraclavicular block with 24C° 20 ml 0,5% bupivacaine
  Interventions: Drug: Bupivacaine Hydrochloride 5 MG/ML
- 37C° 0,5% bupivacaine group (Experimental): 37C° 0,5% bupivacaine group will be performed USG guided infraclavicular block with 37C° 20 ml 0,5% bupivacaine
  Interventions: Drug: Bupivacaine Hydrochloride 5 MG/ML

INTERVENTIONS:
Drug: Bupivacaine Hydrochloride 5 MG/ML — Ultrasound guided infraclavicular brachial plexus block with warmed bupivacaine

SUMMARY:
Brachial plexus blocks have some advantages, but also have some disadvantages as well. As with all nerve blocks, having to wait sometime for an effective block, sometimes failure to achieve an adequate block and possible requirement for isolated nerve block, having to wait a long time for resolution of the block, and immobilization of the extremity for some time can be seen as handicaps for brachial plexus block as well. In the present study, Study was aimed to compare the effects of bupivacaine warmed to body temperature and kept at room temperature on the onset time of ultrasound guided infraclavicular brachial plexus block.

DETAILED DESCRIPTION:
The study design was approved by the locale ethics committee. This double-blinded, randomized, controlled clinical trial recruited 60 patients aged between 18 and 65 years with the American society of anesthesiologists (ASA) physical status classification systems I/II and III who were candidated for surgical operations on any of the forearm, wrist and hand regions. All the participants were asked to sign an informed consent form after having been provided with details of the aim and proceedings of the study.

Patients were excluded from the study if they had a neurological and neuromuscular disorders, psychiatric problems, cardiopulmonary diseases, coagulopathy, infections or allergy to local anesthetic agents.

The patients were equally and randomly distributed into a 24C° 20 ml 0,5% bupivacaine group (Group 1), and 37C° 20 ml 0,5% bupivacaine group (Group 2) via closed envelope technique. All the participants were premedicated with 0.05 mg/kg of intravenous midazolam and monitored routinely before attempting nerve block.

Bupivacaine stored for at least 2 hours in a bain-marie (Memmert Waterbath WNB7, Germany) at 38˚C (regular temperature calibration was made) for Group 2.

The block process was accomplished by an anesthesiologist, who was blind to the temperature of bupivacaine and local anesthetic agent was administered by different anesthesiologist.

At the end of the ICBP block, an anesthetist blinded to the technique evaluated sensory and motor block in every minutes between 5th and 30th minutes as follows. The innervated areas (each dermatome) was evaluated using a pinprick test. The motor block was evaluated by bromage modified scale in every minutes between 10th and 30th minutes. Anxious patients were administered additional midazolam. Subjects refusing awake surgery were administered a propofol infusion with supplemental oxygen as necessary.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged between 18 and 65 years
2. American society of anesthesiologists (ASA) physical status classification systems I/II and III
3. Candidate for surgical operations on any of the forearm, wrist and hand regions.

Exclusion Criteria:

1. Neurological and neuromuscular disorders,
2. Psychiatric problems
3. Cardiopulmonary diseases
4. Coagulopathy
5. Infections
6. Sllergy to local anesthetic agents.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2016-07-01 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
Evaluate sensory block's onset time | 30 minutes after Brachial Plexus Block
  Pain was evaluated by pinprick test (yes-there is a pain/ no-there is no pain)

SECONDARY OUTCOMES:
Evaluate motor block's onset times | 30 minutes after Brachial Plexus Block
  Motion on distal arm was evaluated by bromage scale (0- full flexion of distal arm, 3-unable to move distal arm)

CONTACTS AND LOCATIONS:
Locations (1):
- Palandöken State Hospital, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided